CLINICAL TRIAL: NCT06042348
Title: Placenta Perfusion and Sufficiency Study
Acronym: P2SS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Sahil Joseph Gregory Manoj Sabnani, Principal Investigator, Maxima Medical Center
Other Study IDs: W23.020
Record Dates: First submitted 2023-08-31; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Placenta Diseases, Diagnosis; Pregnancy Related; Female; Human
Keywords: Placenta; Human; Pregnancy; Early pregnancy; Hypertension disorders; Uterus; Uterine artery; Uterine vein; Placental circulation; Placenta physiology; Netherlands; Placenta development
MeSH Terms: conditions — Placenta Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Diagnostic Test: Trans abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: Trans abdominal ultrasound — Ultra sound of the uterus and uterine blood vessels

SUMMARY:
Ultrasonography will be used to determine the total blood flow to and from the uterus. This is done by measuring the blood vessels coming from and going to the uterus. This wil hopefully prove viable and open the possibility to further research in the clinical relevance of these measurements.

DETAILED DESCRIPTION:
This prospective pilot study takes place between 14- and 16-weeks' gestation (GA14 to 16 weeks). This is a feasibility study, as the perfusion measurements have not yet been performed this early in pregnancy. First the feasibility is assessed, before conducting a full-scale research project. The study will take place in a tertiary care obstetric centre, Máxima Medical Center, in Veldhoven The Netherlands. Measurements will be done at the out patient clinic of obstetrics. Duration of the study is 2 months. This gives ample time for recruitment of the subjects.

Recruitment will take place at the outpatient clinic of Máxima Medisch Centrum in Veldhoven. Women with singleton pregnancies coming for their 11-12 weeks' gestational ultrasound, where the pregnancy is dated, will be given a patient information folder in either Dutch or English and asked if the researcher can contact them. Participation is completely on voluntary basis. Patients will be called in the next days by the researcher to answer additional questions and to ask if patients are willing to participate. Contact information of the researchers will be available on the folder in case of questions.

Upon inclusion, the patients will be scheduled for a visit to perform all relevant measurements, henceforth referred to as 'measurement day' (MD) which is to take place between 14- and 16-weeks' gestation. The patient, henceforth to be referred to as participant, will be asked to rest for 5 minutes in a supine position. After 5 minutes of rest the blood pressure of the right arm will be measured, three times using the auto-sphygmomanometer. The three measurements will then be used to calculate the average systolic and diastolic blood pressures. After measurement of blood pressure, the ultrasound scan will be performed. The uterine and placental vessels will be measured according to the standard operating procedure attached to this document. All vessels will be measured 3 times during the ultrasound scan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Between 14-16 weeks gestation on measurement day
* Placenta anterior
* BMI < 30kg/m2
* Ability to give consent
* Adequate mastery of the Dutch or English languages

Exclusion Criteria:

* Non-intact pregnancy at 13 week's gestational echo.
* Vanishing twin
* Multiple gestations
* Congenital or anatomical anomalies at 13 weeks' gestational echo.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The base population are women with singleton pregnancies between 14- and 16 weeks' gestation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Uterine blood vessel flow | Through study completion, an average of 1 year
  The feasibility of measuring placenta perfusion between 14-16 weeks of gestation

SECONDARY OUTCOMES:
uterine vessel differences | Through study completion, an average of 1 year
  To assess whether there are differences in measurements between the two umbilical arteries
Relation between uterine vessels | Through study completion, an average of 1 year
  To determine whether a relation between the uterine artery and vein flow exists

CONTACTS AND LOCATIONS:
Overall Officials: Loes Monen, Principal Investigator — Maxima Medical Center
Locations (1):
- Maxima Medical Center, Veldhoven, Braband, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gude NM, Roberts CT, Kalionis B, King RG. Growth and function of the normal human placenta. Thromb Res. 2004;114(5-6):397-407. doi: 10.1016/j.thromres.2004.06.038. PMID 15507270
- [Background] Fadl S, Moshiri M, Fligner CL, Katz DS, Dighe M. Placental Imaging: Normal Appearance with Review of Pathologic Findings. Radiographics. 2017 May-Jun;37(3):979-998. doi: 10.1148/rg.2017160155. PMID 28493802
- [Background] Brosens I, Pijnenborg R, Vercruysse L, Romero R. The "Great Obstetrical Syndromes" are associated with disorders of deep placentation. Am J Obstet Gynecol. 2011 Mar;204(3):193-201. doi: 10.1016/j.ajog.2010.08.009. Epub 2010 Nov 20. PMID 21094932
- [Background] Schiffer V, van Haren A, De Cubber L, Bons J, Coumans A, van Kuijk SM, Spaanderman M, Al-Nasiry S. Ultrasound evaluation of the placenta in healthy and placental syndrome pregnancies: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2021 Jul;262:45-56. doi: 10.1016/j.ejogrb.2021.04.042. Epub 2021 May 4. PMID 33984727
- [Background] Mol BWJ, Roberts CT, Thangaratinam S, Magee LA, de Groot CJM, Hofmeyr GJ. Pre-eclampsia. Lancet. 2016 Mar 5;387(10022):999-1011. doi: 10.1016/S0140-6736(15)00070-7. Epub 2015 Sep 2. PMID 26342729